CLINICAL TRIAL: NCT01136967
Title: An Open-Label, 2-Cohort, Multicenter, Phase 2 Study of E7080 (Lenvatinib) in Previously Treated Subjects With Unresectable Stage III or Stage IV Melanoma
Brief Title: An Open-Label, 2-Cohort, Multicenter, Study of Lenvatinib in Previously Treated Subjects With Unresectable Stage III or Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7080-G000-206
Record Dates: First submitted 2010-06-02; First posted 2010-06-04 (Estimated); Results first posted 2016-03-16 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2016-11

CONDITIONS: Unresectable Stage III; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (V600E BRAF negative) (Experimental): Cohort 1 (V600E BRAF negative) enrolled participants not harboring the V600E BRAF mutation with disease progression following up to 2 prior systemic anticancer regimens (excluding anti-VEGF) for unresectable Stage III or Stage IV melanoma.
  Interventions: Drug: Lenvatinib
- Cohort 2 (V600E BRAF positive) (Experimental): Cohort 2 (V600E BRAF positive) enrolled participants harboring the activating BRAF mutations (mainly the V600E mutation) with disease progression following BRAF V600E-targeted therapy.
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Participants received lenvatinib 24 mg orally, once daily continuously in 28-day cycles until disease progression, development of unacceptable toxicity or withdrawal of consent.
  Other Names: E7080

SUMMARY:
The purpose of this study is to assess the objective response rate of lenvatinib in previously treated participants with American Joint Committee on Cancer (AJCC) unresectable Stage III or Stage IV melanoma and disease progression.

DETAILED DESCRIPTION:
This was a Phase 2, multicenter, open-label, 2-cohort, 2-stage study that assessed the ORR of lenvatinib in previously treated participants with AJCC unresectable Stage III or Stage IV melanoma and disease progression. Cohort 1 enrolled participants not harboring the V600E BRAF mutation with disease progression following up to 2 prior systemic anticancer regimens (excluding anti-VEGF) for unresectable Stage III or Stage IV melanoma, and is referred to as Cohort 1 or V600E BRAF negative. Other less common BRAF activating mutations were allowed as long as the participant did not receive a BRAF-targeted therapy. Cohort 2 enrolled participants harboring the activating BRAF mutations (mainly the V600E mutation) with disease progression following BRAF V600E-targeted therapy, and is referred to as Cohort 2 or V600E BRAF positive. Eligible participants had measurable disease according to RECIST 1.1.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of melanoma.
2. Unresectable Stage III or Stage IV melanoma.
3. Evidence of disease progression according to RECIST 1.1 on prior regimen.
4. Participants with brain metastases will be eligible if they have undergone complete surgical excision and are more then 1 month post surgery with no radiographic evidence of disease recurrence in the brain or have undergone stereotactic radio surgery (gamma knife procedure) and are more then 1 month post procedure and with no radiographic evidence of disease progression in the brain; and are asymptomatic, and discontinued corticosteroid treatment at least 30 days prior starting treatment.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Adequately controlled blood pressure.
7. Adequate renal function, bone marrow function, blood coagulation function, and liver function, as defined in the study protocol.

Exclusion Criteria:

1. Melanoma of intraocular origin.
2. Leptomeningeal metastases or brain metastases except as for participants with brain metastases will be eligible if they have undergone complete surgical excision and are more then 1 month post surgery with no radiographic evidence of disease recurrence in the brain or have undergone stereotactic radio surgery (gamma knife procedure) and are more then 1 month post procedure and with no radiographic evidence of disease progression in the brain; and are asymptomatic, and discontinued corticosteroid treatment at least 30 days prior starting treatment.
3. More than 2 prior systemic anticancer regimen treatments including immunotherapies for unresectable Stage III or Stage IV disease (if BRAF V600E mutation negative) or not previously treated with BRAF V600E-targeted therapy or received in the past more than 2 prior systemic anticancer regimen treatments, including immunotherapies, in addition to a BRAF-V600E-targeted therapy (if BRAF V600E mutation positive).
4. Significant cardiovascular impairment.
5. Bleeding disorder or a thrombotic disorder requiring anticoagulant therapy.
6. Females who are pregnant or breastfeeding.
7. Prolongation of QTc interval to greater than 480 msec.
8. 24 hour urine protein greater than or equal to 1 gm.
9. Active hemoptysis within 3 wks prior to the first dose of study drug.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eisai US Medical Services, Study Director — Eisai Limited
Locations (95):
- United States (79):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Los Angeles, California
  - San Francisco, California
  - Aurora, Colorado
  - Boulder, Colorado
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Lakewood, Colorado
  - Littleton, Colorado
  - Lone Tree, Colorado
  - Longmont, Colorado
  - Parker, Colorado
  - Thornton, Colorado
  - Bonita Springs, Florida
  - Bradenton, Florida
  - Cape Coral, Florida
  - Clearwater, Florida
  - Englewood, Florida
  - Fort Myers, Florida
  - Gainesville, Florida
  - Naples, Florida
  - North Port, Florida
  - Orlando, Florida
  - Palm Harbor, Florida
  - Port Charlotte, Florida
  - Sarasota, Florida
  - Sebring, Florida
  - Tampa, Florida
  - Venice, Florida
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Detroit, Michigan
  - Burnsville, Minnesota
  - Coon Rapids, Minnesota
  - Edina, Minnesota
  - Fridley, Minnesota
  - Maplewood, Minnesota
  - Minneapolis, Minnesota
  - Saint Paul, Minnesota
  - Woodbury, Minnesota
  - Southaven, Mississippi
  - St Louis, Missouri
  - Henderson, Nevada
  - Las Vegas, Nevada
  - Lebanon, New Hampshire
  - Morristown, New Jersey
  - New York, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Eugene, Oregon
  - Portland, Oregon
  - Springfield, Oregon
  - Tualatin, Oregon
  - Bethlehem, Pennsylvania
  - Philadelphia, Pennsylvania
  - Bartlett, Tennessee
  - Franklin, Tennessee
  - Gallatin, Tennessee
  - Germantown, Tennessee
  - Hermitage, Tennessee
  - Lebanon, Tennessee
  - Memphis, Tennessee
  - Murfreesboro, Tennessee
  - Nashville, Tennessee
  - Smyrna, Tennessee
  - Bedford, Texas
  - Dallas, Texas
  - Grapevine, Texas
  - Houston, Texas
  - Arlington, Virginia
  - Fairfax, Virginia
  - Gainesville, Virginia
  - Leesburg, Virginia
  - Winchester, Virginia
  - Woodbridge, Virginia
  - Vancouver, Washington
  - Madison, Wisconsin
- Australia (6):
  - Adelaide
  - Malvern
  - Newcastle
  - North Sydney
  - Perth
  - Westmead
- Germany (6):
  - Essen
  - Hanover
  - Heidelberg
  - Kiel
  - Mainz
  - Tübingen
- United Kingdom (4):
  - Glasgow
  - London
  - Nottingham
  - Surrey

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 298 participants were screened. Of these, 116 were screen failures and 182 received treatment (93 participants in Cohort 1 and 89 participants in Cohort 2).
Groups:
- Cohort 1 (V600E BRAF Negative): Cohort 1 (V600E BRAF negative) enrolled participants not harboring the V600E BRAF mutation with disease progression following up to 2 prior systemic anticancer regimens (excluding anti-VEGF) for unresectable Stage III or Stage IV melanoma. Participants received lenvatinib 24 mg orally, once daily continuously in 28-day cycles.
- Cohort 2 (V600E BRAF Positive): Cohort 2 (V600E BRAF positive) enrolled participants harboring the activating BRAF mutations (mainly the V600E mutation) with disease progression following BRAF V600E-targeted therapy. Participants received lenvatinib 24 mg orally, once daily continuously in 28-day cycles.
Period: Overall Study
Arm/Group | Cohort 1 (V600E BRAF Negative) | Cohort 2 (V600E BRAF Positive)
Started | 93 | 89
Disease Progression | 55 | 56
Treatment Ongoing at Data Cutoff | 14 (Entered Extension Phase on treatment at data cut-off (18 January 2012)) | 6 (Entered Extension Phase on treatment at data cut-off (15 April 2013))
Completed | 69 (Disease Progression and treatment ongoing at data cutoff (18 January 2012)) | 62 (Disease Progression and treatment ongoing at data cutoff (15 April 2013))
Not Completed | 24 | 27
Not completed — Adverse Event | 9 | 12
Not completed — Participant Choice | 8 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Clinical Progression | 3 | 5
Not completed — Radiation | 1 | 0
Not completed — Non-compliance | 1 | 0
Not completed — Investigator's Choice | 1 | 1
Not completed — Increase in Lesion Size | 0 | 2
Not completed — Diagnosis of Second Primary Cancer | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (V600E BRAF Negative) | Cohort 2 (V600E BRAF Positive) | Total
Number analyzed (Participants) | 93 | 89 | 182
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.5 (11.71) | 55.0 (14.18) | 58.8 (13.47)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 29 | 39 | 68
  Male | 64 | 50 | 114
AJCC Melanoma Tumor, Node, Metastasis (TNM) Stage at Study Entry [Number; unit: Participants] — American joint committee on cancer (AJCC) (8th edition) staging system for melanoma tumor categorize the tumor in five stages: Stage 0: no evidence of primary tumor/early cancer that has not spread to neighboring tissue; Stage 1: tumor thickness measurements less than or equal to (<=)1.0 millimeter (mm); Stage 2: tumor thickness measurements greater than (>)1.0 mm to 2.0 mm; Stage 3: tumor thickness measurements >2.0 mm to 4.0 mm; Stage 4: tumor thickness measurements >4.0 mm. Higher stage of tumor shows worse outcomes.
  Participants
    Unresectable Stage III | 5 | 7 | 12
    Unresectable Stage IV | 88 | 82 | 170

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR, (ORR = CR + PR) was defined as the percentage of participants in each cohort who had a best overall response (BOR) of complete response (CR) or partial response (PR) based on Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 for target lesions assessed by magnetic resonance imaging/computed tomography (MRI/CT) scans and independent radiologic review (IRR). A BOR of CR required confirmation by a subsequent CR assessment at least 4 weeks later. A BOR of PR required confirmation by a subsequent assessment of CR or PR at least 4 weeks later. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (target or non-target) had to have a reduction in short axis to less than (<)10 mm. PR was defined as at least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of treatment start until all participants completed a minimum of 6 cycles (28-day cycles) or discontinued treatment prior to end of Cycle 6 (up to 24 weeks)
Population: Full Analysis Set (Intent-to-Treat [ITT] Analysis Set) included all participants who received at least 1 dose study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1 (V600E BRAF Negative) | Cohort 2 (V600E BRAF Positive)
Number analyzed (Participants) | 93 | 89
Percentage of participants | 8.6 [3.8 to 16.2] | 9.0 [4.0 to 16.9]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was measured as the time from the date of first administration of study treatment until the date of first documentation of disease progression or date of death from any cause (whichever occurred first), as determined by IRR and Investigator based on RECIST v1.1. Disease progression per RECIST v1.1 was defined as at least a 20% relative increase and 5 mm absolute increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) recorded since the treatment started or the appearance of 1 or more new lesions. PFS was analyzed using Kaplan-Meier (1958) product-limit estimates. Data were presented with 2-sided 95% confidence interval (CI) when an adequate number of at risk participants warranted the estimates in the table below.
Time Frame: From date of treatment start until documentation of disease progression or death from any cause (whichever occurred first) or up to data cutoff (Cohort 1; 15 Jan 2012 and Cohort 2; 15 Apr 2013), up to approximately 2 years 8 months
Population: Full Analysis Set (ITT Analysis Set) included all participants who received at least 1 dose study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 (V600E BRAF Negative) | Cohort 2 (V600E BRAF Positive)
Number analyzed (Participants) | 93 | 89
Months
  Determined by IRR | 3.7 [2.5 to 4.2] | 1.8 [1.8 to 2.2]
  Determined by Investigator | 3.7 [3.6 to 4.2] | 2.3 [1.9 to 3.4]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the length of time in months from the date of first administration of study drug until the date of death from any cause, and was based on the data cutoff date for each cohort. OS was analyzed using Kaplan-Meier (1958) product-limit estimates. Data were presented with 2-sided 95% CI when an adequate number of at risk participants warranted the estimates in the table below.
Time Frame: From date of treatment start until date of death from any cause or up to data cutoff (Cohort 1; 15 Jan 2012 and Cohort 2; 15 Apr 2013), up to approximately 2 years 8 months
Population: Full Analysis Set (ITT Analysis Set) included all participants who received at least 1 dose study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 (V600E BRAF Negative) | Cohort 2 (V600E BRAF Positive)
Number analyzed (Participants) | 93 | 89
Months | 8.9 [8.3 to NA] — NA: Not applicable since the upper limit of the 95% confidence interval was not yet reached at the time of analysis. | 6.3 [5.2 to 8.8]

4. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR, (DCR = CR + PR + SD) was defined as the percentage of participants who had a BOR of CR or PR or stable disease (SD) based on RECIST v1.1 for target lesions assessed by MRI/CT and IRR. CR was defined as the disappearance of all target lesions, any pathological lymph nodes (target or non-target) had to have a reduction in short axis to <10 mm.; PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; Overall Response (OR) = CR + PR. SD defined as reduction in tumor volume of < 30% or an increase in the volume of 1 or more measurable lesions of < 25% without the appearance of any new lesions which was neither tumor shrinkage corresponding to PR nor tumor expansion corresponding to disease progression. BOR of SD, time from first administration of study drug until date of documented SD needed to be >=7 weeks based on IRR and Investigator's assessment.
Time Frame: as for outcome 2
Population: Full Analysis Set (ITT Analysis Set) included all participants who received at least 1 dose study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1 (V600E BRAF Negative) | Cohort 2 (V600E BRAF Positive)
Number analyzed (Participants) | 93 | 89
Percentage of participants
  Determined by IRR | 52.7 [42.1 to 63.1] | 34.8 [25.0 to 45.7]
  Determined by Investigator | 64.5 [53.9 to 74.2] | 48.3 [37.6 to 59.2]

5. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR, (CBR = CR + PR + durable SD rate) was defined as the percentage of participants who had a BOR of CR or PR or durable SD (dSD, SD lasting >=23 weeks) based on RECIST v1.1 for target lesions assessed by MRI/CT, IRR and Investigator's assessment. A BOR of CR required confirmation by a subsequent CR assessment at least 4 weeks later. A BOR of PR required confirmation by a subsequent assessment of CR or PR at least 4 weeks later. CR was defined as the disappearance of all target lesions, any pathological lymph nodes (target or non-target) had to have a reduction in short axis to less than 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; OR = CR + PR. A BOR of dSD, the time from the first administration of study drug until the date of documented dSD needed to be ≥23 weeks based on IRR and Investigator's assessment.
Time Frame: as for outcome 2
Population: Full Analysis Set (ITT Analysis Set) included all participants who received at least 1 dose study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1 (V600E BRAF Negative) | Cohort 2 (V600E BRAF Positive)
Number analyzed (Participants) | 93 | 89
Percentage of participants
  Determined by IRR | 31.2 [22.0 to 41.6] | 14.6 [8.0 to 23.7]
  Determined by Investigator | 33.3 [23.9 to 43.9] | 20.2 [12.4 to 30.1]

6. Secondary Outcome: Number of Participants With Adverse Events (AEs)/ Serious Adverse Events (SAEs) as a Measure of Safety and Tolerability of Lenvatinib
Description: Safety was assessed by monitoring and recording all AEs including all Common Terminology Criteria for Adverse Events (CTCAE) grades and SAEs; regular monitoring of hematology, clinical chemistry, and urine values; physical examinations; and regular measurement of vital signs, electrocardiograms (ECGs), and multi-gated acquisition (MUGA) scans or echocardiogram.
Time Frame: From date of treatment start up to 30 days after the last dose, or up to data cutoff (Cohort 1; 15 Jan 2012 and Cohort 2; 15 Apr 2013), up to approximately 2 years 9 months
Population: Safety Analysis Set included those participants who received at least 1 dose of study drug and had at least 1 post baseline safety evaluation.
Measure: Number; unit: Participants
Arm/Group | Cohort 1 (V600E BRAF Negative) | Cohort 2 (V600E BRAF Positive)
Number analyzed (Participants) | 93 | 89
Participants
  AEs | 93 | 89
  SAEs | 39 | 36

7. Secondary Outcome: Change From Baseline in the Concentration of Clinical Biomarkers in Whole Blood
Description: Blood samples were drawn at specific time points. Utilizing a standard protocol, the deoxyribonucleic acid (DNA) from whole blood was extracted and analyzed for specific biomarkers of absorption, distribution, metabolism, and excretion of lenvatinib. Some of the biomarkers analyzed included; Angiopoietin, Epidermal Growth Factor (EGF), Fibroblast Growth Factor (FGF), FMS Like Tyrosine Kinase 3 Ligand (Flt3l) Granulocyte Colony Stimulating Factor (G-CSF), Granulocyte Macro Colony Stimulating Factor (GM-CSF), Interleukin 1 Receptor Antagonist (IL-1RA), Interferon (IFN), Macrophage Inflammatory Protein (MIP) 1 alpha, Platelet Derived Growth Factor (PDGF), Stromal Cell Derived Factor (SDF) 1 alpha, Interleukin (IL), Transforming Growth Factor (TGF), Tumor Necrosis Factor (TNF), Vascular Endothelial Growth Factor (VEGF).
Time Frame: Cycle 1 Day 15 (C1 D15), Cycle 2 Day 1 (C2 D1), Cycle 3 Day 1 (C3 D1), Off-Treatment/Phase Visit 98 (V98)
Population: The Safety Analysis set was used and included all participants who received at least one dose of lenvatinib and had at least 1 postbaseline safety evaluation. Number analyzed (n) signifies participants who were evaluable at specific time points for this outcome measure.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cohort 1 (V600E BRAF Negative) | Cohort 2 (V600E BRAF Positive)
Number analyzed (Participants) | 93 | 89
pg/mL
  Angiopoietin 2 76 C1D15: number analyzed (Participants) | 78 | 0
  Angiopoietin 2 76 C1D15 | -1015.69 (946.596) |
  Angiopoietin 2 76 C2D1: number analyzed (Participants) | 79 | 0
  Angiopoietin 2 76 C2D1 | -832.29 (1257.287) |
  Angiopoietin 2 76 C3D1: number analyzed (Participants) | 51 | 0
  Angiopoietin 2 76 C3D1 | -923.82 (969.285) |
  Angiopoietin 2 76 V98: number analyzed (Participants) | 6 | 0
  Angiopoietin 2 76 V98 | -947.00 (825.037) |
  Angiopoietin 2 90 C1D15: number analyzed (Participants) | 0 | 69
  Angiopoietin 2 90 C1D15 |  | -1225.322 (1950.4525)
  Angiopoietin 2 90 C2D1: number analyzed (Participants) | 0 | 66
  Angiopoietin 2 90 C2D1 |  | -1100.235 (1378.4621)
  Angiopoietin 2 90 C3D1: number analyzed (Participants) | 0 | 0
  Angiopoietin 2 90 V98: number analyzed (Participants) | 0 | 0
  Angiopoietin 1 C1D15: number analyzed (Participants) | 80 | 70
  Angiopoietin 1 C1D15 | -3033.030 (8808.2059) | -2717.533 (16689.4536)
  Angiopoietin 1 C2D1: number analyzed (Participants) | 80 | 67
  Angiopoietin 1 C2D1 | -2802.306 (10202.7814) | -1743.569 (15546.4804)
  Angiopoietin 1 C3D1: number analyzed (Participants) | 52 | 0
  Angiopoietin 1 C3D1 | -859.021 (9994.6711) |
  Angiopoietin 1 V98: number analyzed (Participants) | 6 | 0
  Angiopoietin 1 V98 | 8107.400 (17740.0516) |
  Angiopoietin 2 C1D15: number analyzed (Participants) | 80 | 70
  Angiopoietin 2 C1D15 | -1462.552 (1541.8074) | -2154.269 (3560.0029)
  Angiopoietin 2 C2D1: number analyzed (Participants) | 80 | 67
  Angiopoietin 2 C2D1 | -1225.462 (1872.5841) | -1884.439 (2357.1979)
  Angiopoietin 2 C3D1: number analyzed (Participants) | 52 | 0
  Angiopoietin 2 C3D1 | -1255.485 (1738.0891) |
  Angiopoietin 2 V98: number analyzed (Participants) | 6 | 0
  Angiopoietin 2 V98 | -1374.183 (1158.2897) |
  CD40 Ligand C1D15: number analyzed (Participants) | 59 | 70
  CD40 Ligand C1D15 | -24020.778 (62788.2464) | -4678.661 (41191.7303)
  CD40 Ligand C2D1: number analyzed (Participants) | 58 | 67
  CD40 Ligand C2D1 | -22957.613 (73677.4378) | -7254.754 (37794.5541)
  CD40 Ligand C3D1: number analyzed (Participants) | 35 | 0
  CD40 Ligand C3D1 | -16700.900 (48016.0710) |
  CD40 Ligand V98: number analyzed (Participants) | 3 | 0
  CD40 Ligand V98 | 2192.177 (86909.9688) |
  EGF 2 C1D15: number analyzed (Participants) | 74 | 62
  EGF 2 C1D15 | -46.493 (101.0772) | -0.516 (219.9787)
  EGF 2 C2D1: number analyzed (Participants) | 76 | 58
  EGF 2 C2D1 | -39.636 (125.0664) | -29.803 (121.1705)
  EGF 2 C3D1: number analyzed (Participants) | 47 | 0
  EGF 2 C3D1 | -37.600 (113.8543) |
  EGF 2 V98: number analyzed (Participants) | 6 | 0
  EGF 2 V98 | -2.230 (191.4129) |
  EGF 59 C1D15: number analyzed (Participants) | 77 | 0
  EGF 59 C1D15 | -37.07 (81.051) |
  EGF 59 C2D1: number analyzed (Participants) | 78 | 0
  EGF 59 C2D1 | -31.58 (96.200) |
  EGF 59 C3D1: number analyzed (Participants) | 50 | 0
  EGF 59 C3D1 | -24.49 (93.102) |
  EGF 59 V98: number analyzed (Participants) | 6 | 0
  EGF 59 V98 | 10.17 (137.755) |
  EGF 80 C1D15: number analyzed (Participants) | 0 | 65
  EGF 80 C1D15 |  | -31.519 (126.2579)
  EGF 80 C2D1: number analyzed (Participants) | 0 | 65
  EGF 80 C2D1 |  | -32.171 (121.7805)
  EGF 80 C3D1: number analyzed (Participants) | 0 | 0
  EGF 80 V98: number analyzed (Participants) | 0 | 0
  Eotaxin-4 C1D15: number analyzed (Participants) | 78 | 70
  Eotaxin-4 C1D15 | 51.456 (117.1266) | 46.538 (128.398)
  Eotaxin-4 C2D1: number analyzed (Participants) | 79 | 67
  Eotaxin-4 C2D1 | 99.974 (207.0243) | 60.919 (114.6134)
  Eotaxin-4 C3D1: number analyzed (Participants) | 50 | 0
  Eotaxin-4 C3D1 | 89.878 (108.6392) |
  Eotaxin-4 V98: number analyzed (Participants) | 6 | 0
  Eotaxin-4 V98 | 104.613 (157.7527) |
  FGF 2 C1D15: number analyzed (Participants) | 77 | 57
  FGF 2 C1D15 | -4.294 (51.3985) | 8.325 (136.3433)
  FGF 2 C2D1: number analyzed (Participants) | 78 | 54
  FGF 2 C2D1 | -8.085 (48.8273) | -8.003 (144.9054)
  FGF 2 C3D1: number analyzed (Participants) | 51 | 0
  FGF 2 C3D1 | 7.443 (45.7310) |
  FGF 2 V98: number analyzed (Participants) | 6 | 0
  FGF 2 V98 | -3.917 (62.3623) |
  FGF 23 C1D15: number analyzed (Participants) | 32 | 0
  FGF 23 C1D15 | 6.549 (22.5297) |
  FGF 23 C2D1: number analyzed (Participants) | 36 | 0
  FGF 23 C2D1 | 6.496 (27.2305) |
  FGF 23 C3D1: number analyzed (Participants) | 22 | 0
  FGF 23 C3D1 | 6.691 (24.5203) |
  FGF 23 V98: number analyzed (Participants) | 2 | 0
  FGF 23 V98 | 13.430 (36.7130) |
  FGF 4 C1D15: number analyzed (Participants) | 68 | 25
  FGF 4 C1D15 | -24.226 (100.6823) | 50.369 (253.9626)
  FGF 4 C2D1: number analyzed (Participants) | 68 | 23
  FGF 4 C2D1 | -15.491 (104.9991) | 55.785 (264.4585)
  FGF 4 C3D1: number analyzed (Participants) | 47 | 0
  FGF 4 C3D1 | 5.283 (130.3452) |
  FGF 4 V98: number analyzed (Participants) | 5 | 0
  FGF 4 V98 | 33.860 (185.4616) |
  FGF Basic Form C1D15: number analyzed (Participants) | 68 | 44
  FGF Basic Form C1D15 | -0.597 (18.6851) | 43.457 (224.9856)
  FGF Basic Form C2D1: number analyzed (Participants) | 68 | 41
  FGF Basic Form C2D1 | -1.212 (38.4131) | 64.237 (328.6676)
  FGF Basic Form C3D1: number analyzed (Participants) | 44 | 0
  FGF Basic Form C3D1 | 2.060 (29.2405) |
  FGF Basic Form V98: number analyzed (Participants) | 5 | 0
  FGF Basic Form V98 | 18.384 (28.6214) |
  Flt3l C1D15: number analyzed (Participants) | 78 | 69
  Flt3l C1D15 | -0.037 (32.5371) | -8.877 (23.0368)
  Flt3l C2D1: number analyzed (Participants) | 79 | 66
  Flt3l C2D1 | 5.135 (28.0359) | -1.362 (39.2251)
  Flt3l C3D1: number analyzed (Participants) | 51 | 0
  Flt3l C3D1 | 5.439 (24.1985) |
  Flt3l V98: number analyzed (Participants) | 6 | 0
  Flt3l V98 | 13.367 (17.7279) |
  Fractalkine C1D15: number analyzed (Participants) | 68 | 56
  Fractalkine C1D15 | -11.700 (94.5115) | 38.670 (237.5045)
  Fractalkine C2D1: number analyzed (Participants) | 69 | 54
  Fractalkine C2D1 | -1.175 (70.0858) | 4.663 (58.1950)
  Fractalkine C3D1: number analyzed (Participants) | 47 | 0
  Fractalkine C3D1 | -5.588 (116.3955) |
  Fractalkine V98: number analyzed (Participants) | 4 | 0
  Fractalkine V98 | 15.838 (90.6004) |
  G-CSF C1D15: number analyzed (Participants) | 78 | 70
  G-CSF C1D15 | 4.329 (20.8343) | 6.368 (61.7181)
  G-CSF C2D1: number analyzed (Participants) | 79 | 66
  G-CSF C2D1 | 7.366 (32.5552) | 12.601 (72.5113)
  G-CSF C3D1: number analyzed (Participants) | 50 | 0
  G-CSF C3D1 | 11.292 (24.1828) |
  G-CSF V98: number analyzed (Participants) | 6 | 0
  G-CSF V98 | 34.653 (101.7055) |
  GM-CSF C1D15: number analyzed (Participants) | 36 | 26
  GM-CSF C1D15 | 0.767 (16.9314) | 44.665 (220.9124)
  GM-CSF C2D1: number analyzed (Participants) | 42 | 27
  GM-CSF C2D1 | 4.371 (38.3355) | 139.491 (725.0903)
  GM-CSF C3D1: number analyzed (Participants) | 29 | 0
  GM-CSF C3D1 | 10.036 (49.8538) |
  GM-CSF V98: number analyzed (Participants) | 2 | 0
  GM-CSF V98 | -1.495 (5.1831) |
  Growth Regulated Oncogene C1D15: number analyzed (Participants) | 0 | 70
  Growth Regulated Oncogene C1D15 |  | -141.838 (410.3579)
  Growth Regulated Oncogene C2D1: number analyzed (Participants) | 0 | 67
  Growth Regulated Oncogene C2D1 |  | -120.148 (456.3073)
  Growth regulated oncogene C3D1: number analyzed (Participants) | 0 | 0
  Growth regulated oncogene V98: number analyzed (Participants) | 0 | 0
  Hepatocyte Growth Factor C1D15: number analyzed (Participants) | 78 | 68
  Hepatocyte Growth Factor C1D15 | 102.527 (1309.4077) | -91.790 (781.2225)
  Hepatocyte Growth Factor C2D1: number analyzed (Participants) | 78 | 65
  Hepatocyte Growth Factor C2D1 | -126.667 (693.2257) | -147.796 (411.1836)
  Hepatocyte Growth Factor C3D1: number analyzed (Participants) | 51 | 0
  Hepatocyte Growth Factor C3D1 | 61.257 (1062.3266) |
  Hepatocyte Growth Factor V98: number analyzed (Participants) | 6 | 0
  Hepatocyte Growth Factor V98 | 404.700 (456.8130) |
  Interferon Gamma C1D15: number analyzed (Participants) | 31 | 18
  Interferon Gamma C1D15 | 4.072 (19.3994) | 33.743 (100.3678)
  Interferon Gamma C2D1: number analyzed (Participants) | 32 | 18
  Interferon Gamma C2D1 | -0.392 (14.8083) | -10.164 (170.9869)
  Interferon Gamma C3D1: number analyzed (Participants) | 21 | 0
  Interferon Gamma C3D1 | 2.986 (5.7591) |
  Interferon Gamma V98: number analyzed (Participants) | 2 | 0
  Interferon Gamma V98 | 2.455 (5.2255) |
  Interleukin 1 alpha C1D15: number analyzed (Participants) | 25 | 16
  Interleukin 1 alpha C1D15 | 0.159 (7.9441) | 67.203 (200.9806)
  Interleukin 1 alpha C2D1: number analyzed (Participants) | 28 | 16
  Interleukin 1 alpha C2D1 | 0.226 (8.2728) | -36.352 (198.1416)
  Interleukin 1 alpha C3D1: number analyzed (Participants) | 22 | 0
  Interleukin 1 alpha C3D1 | -0.140 (13.7136) |
  Interleukin 1 alpha V98: number analyzed (Participants) | 0 | 0
  Interleukin 1 Beta C1D15: number analyzed (Participants) | 16 | 6
  Interleukin 1 Beta C1D15 | 0.279 (1.9668) | 59.768 (137.6657)
  Interleukin 1 Beta C2D1: number analyzed (Participants) | 19 | 6
  Interleukin 1 Beta C2D1 | 1.198 (5.0044) | 27.690 (61.2456)
  Interleukin 1 Beta C3D1: number analyzed (Participants) | 13 | 0
  Interleukin 1 Beta C3D1 | 1.882 (11.1737) |
  Interleukin 1 Beta V98: number analyzed (Participants) | 0 | 0
  IL-1RA C1D15: number analyzed (Participants) | 40 | 18
  IL-1RA C1D15 | 14.490 (63.5869) | 46.381 (132.3985)
  IL-1RA C2D1: number analyzed (Participants) | 43 | 16
  IL-1RA C2D1 | 20.295 (61.9799) | 38.131 (142.7521)
  IL-1RA C3D1: number analyzed (Participants) | 29 | 0
  IL-1RA C3D1 | 7.048 (30.9383) |
  IL-1RA V98: number analyzed (Participants) | 5 | 0
  IL-1RA V98 | 84.614 (178.1590) |
  Interleukin 12 (p40) C1D15: number analyzed (Participants) | 45 | 19
  Interleukin 12 (p40) C1D15 | 14.514 (73.9806) | 5.458 (28.8514)
  Interleukin 12 (p40) C2D1: number analyzed (Participants) | 49 | 19
  Interleukin 12 (p40) C2D1 | 16.052 (40.3849) | 918.03 (3917.8689)
  Interleukin 12 (p40) C3D1: number analyzed (Participants) | 35 | 0
  Interleukin 12 (p40) C3D1 | 11.183 (36.3506) |
  Interleukin 12 (p40) V98: number analyzed (Participants) | 2 | 0
  Interleukin 12 (p40) V98 | -8.130 (5.7276) |
  Interleukin 12 (p70) C1D15: number analyzed (Participants) | 17 | 14
  Interleukin 12 (p70) C1D15 | 1.241 (18.8429) | 27.919 (62.8944)
  Interleukin 12 (p70) C2D1: number analyzed (Participants) | 21 | 14
  Interleukin 12 (p70) C2D1 | -5.622 (28.6381) | 7.820 (71.1505)
  Interleukin 12 (p70) C3D1: number analyzed (Participants) | 15 | 0
  Interleukin 12 (p70) C3D1 | -6.099 (19.5015) |
  Interleukin 12 (p70) V98: number analyzed (Participants) | 2 | 0
  Interleukin 12 (p70) V98 | 11.275 (20.0182) |
  Interleukin 10 C1D15: number analyzed (Participants) | 34 | 40
  Interleukin 10 C1D15 | -5.170 (38.0092) | -7.611 (22.1926)
  Interleukin 10 C2D1: number analyzed (Participants) | 37 | 41
  Interleukin 10 C2D1 | -1.901 (33.6203) | 1.687 (72.7629)
  Interleukin 10 C3D1: number analyzed (Participants) | 22 | 0
  Interleukin 10 C3D1 | 4.136 (10.8185) |
  Interleukin 10 V98: number analyzed (Participants) | 2 | 0
  Interleukin 10 V98 | -28.065 (41.7547) |
  Interleukin 13 C1D15: number analyzed (Participants) | 22 | 5
  Interleukin 13 C1D15 | 0.961 (5.0066) | 8.574 (13.4754)
  Interleukin 13 C2D1: number analyzed (Participants) | 23 | 5
  Interleukin 13 C2D1 | 2.451 (7.6374) | 8.536 (18.5220)
  Interleukin 13 C3D1: number analyzed (Participants) | 17 | 0
  Interleukin 13 C3D1 | 5.404 (16.4719) |
  Interleukin 13 V98: number analyzed (Participants) | 0 | 0
  Interleukin 15 C1D15: number analyzed (Participants) | 21 | 8
  Interleukin 15 C1D15 | 0.128 (2.2957) | 85.619 (234.7106)
  Interleukin 15 C2D1: number analyzed (Participants) | 23 | 9
  Interleukin 15 C2D1 | 1.403 (4.1630) | 574.776 (1709.9272)
  Interleukin 15 C3D1: number analyzed (Participants) | 16 | 0
  Interleukin 15 C3D1 | -0.178 (3.6993) |
  Interleukin 15 V98: number analyzed (Participants) | 1 | 0
  Interleukin 15 V98 | 3.930 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. |
  Interleukin 17 C1D15: number analyzed (Participants) | 24 | 9
  Interleukin 17 C1D15 | 3.434 (8.6463) | 4.567 (12.1008)
  Interleukin 17 C2D1: number analyzed (Participants) | 24 | 11
  Interleukin 17 C2D1 | 1.264 (8.0963) | 3.035 (15.8736)
  Interleukin 17 C3D1: number analyzed (Participants) | 15 | 0
  Interleukin 17 C3D1 | 0.011 (3.4100) |
  Interleukin 17 V98: number analyzed (Participants) | 2 | 0
  Interleukin 17 V98 | 8.440 (11.7663) |
  Interleukin 2 C1D15: number analyzed (Participants) | 14 | 6
  Interleukin 2 C1D15 | -1.004 (7.1024) | 173.878 (397.2754)
  Interleukin 2 C2D1: number analyzed (Participants) | 9 | 6
  Interleukin 2 C2D1 | 5.853 (20.3294) | 191.410 (461.1991)
  Interleukin 2 C3D1: number analyzed (Participants) | 11 | 0
  Interleukin 2 C3D1 | 2.647 (19.5979) |
  Interleukin 2 V98: number analyzed (Participants) | 0 | 0
  Interleukin 4 C1D15: number analyzed (Participants) | 23 | 39
  Interleukin 4 C1D15 | 8.169 (30.0305) | 12.815 (77.4310)
  Interleukin 4 C2D1: number analyzed (Participants) | 23 | 40
  Interleukin 4 C2D1 | 20.167 (77.0619) | 7.815 (54.5735)
  Interleukin 4 C3D1: number analyzed (Participants) | 20 | 0
  Interleukin 4 C3D1 | 6.583 (20.3824) |
  Interleukin 4 V98: number analyzed (Participants) | 0 | 0
  Interleukin 5 C1D15: number analyzed (Participants) | 9 | 5
  Interleukin 5 C1D15 | 0.311 (1.1314) | 6.088 (7.5239)
  Interleukin 5 C2D1: number analyzed (Participants) | 10 | 6
  Interleukin 5 C2D1 | 0.205 (1.5931) | 11.382 (9.8663)
  Interleukin 5 C3D1: number analyzed (Participants) | 6 | 0
  Interleukin 5 C3D1 | -0.327 (1.1102) |
  Interleukin 5 V98: number analyzed (Participants) | 0 | 0
  Interleukin 6 C1D15: number analyzed (Participants) | 35 | 39
  Interleukin 6 C1D15 | 0.166 (6.8774) | 3.784 (30.0715)
  Interleukin 6 C2D1: number analyzed (Participants) | 34 | 36
  Interleukin 6 C2D1 | 4.778 (34.0254) | 5.524 (32.1205)
  Interleukin 6 C3D1: number analyzed (Participants) | 21 | 0
  Interleukin 6 C3D1 | 2.027 (7.3121) |
  Interleukin 6 V98: number analyzed (Participants) | 4 | 0
  Interleukin 6 V98 | 3.160 (6.6276) |
  Interleukin 7 C1D15: number analyzed (Participants) | 26 | 20
  Interleukin 7 C1D15 | 1.267 (7.3732) | 2.167 (8.8122)
  Interleukin 7 C2D1: number analyzed (Participants) | 28 | 21
  Interleukin 7 C2D1 | 2.413 (8.8367) | 5.744 (18.4339)
  Interleukin 7 C3D1: number analyzed (Participants) | 19 | 0
  Interleukin 7 C3D1 | 0.616 (5.0590) |
  Interleukin 7 V98: number analyzed (Participants) | 2 | 0
  Interleukin 7 V98 | 20.760 (28.0439) |
  Interleukin 8 C1D15: number analyzed (Participants) | 78 | 68
  Interleukin 8 C1D15 | -5.801 (46.1572) | -20.769 (52.1135)
  Interleukin 8 C2D1: number analyzed (Participants) | 79 | 65
  Interleukin 8 C2D1 | -5.431 (43.4197) | -14.303 (57.9561)
  Interleukin 8 C3D1: number analyzed (Participants) | 50 | 0
  Interleukin 8 C3D1 | -7.348 (43.0509) |
  Interleukin 8 V98: number analyzed (Participants) | 6 | 0
  Interleukin 8 V98 | 26.982 (32.7795) |
  IFN gamma Induced Protein 10 C1D15: number analyzed (Participants) | 78 | 70
  IFN gamma Induced Protein 10 C1D15 | 453.684 (1446.5825) | 184.891 (501.5782)
  IFN gamma Induced Protein 10 C2D1: number analyzed (Participants) | 79 | 67
  IFN gamma Induced Protein 10 C2D1 | 246.194 (246.194) | 306.075 (792.5621)
  IFN gamma Induced Protein 10 C3D1: number analyzed (Participants) | 50 | 0
  IFN gamma Induced Protein 10 C3D1 | 201.923 (483.5088) |
  IFN gamma Induced Protein 10 V98: number analyzed (Participants) | 6 | 0
  IFN gamma Induced Protein 10 V98 | 359.872 (501.1082) |
  Monocyte Chemotactic Protein 1 C1D15: number analyzed (Participants) | 78 | 70
  Monocyte Chemotactic Protein 1 C1D15 | 0.733 (423.2721) | -101.580 (371.5381)
  Monocyte Chemotactic Protein 1 C2D1: number analyzed (Participants) | 79 | 67
  Monocyte Chemotactic Protein 1 C2D1 | -19.036 (372.5242) | 128.749 (541.1034)
  Monocyte Chemotactic Protein 1 C3D1: number analyzed (Participants) | 50 | 0
  Monocyte Chemotactic Protein 1 C3D1 | 13.542 (370.3700) |
  Monocyte Chemotactic Protein 1 V98: number analyzed (Participants) | 6 | 0
  Monocyte Chemotactic Protein 1 V98 | -128.627 (1234.5888) |
  MIP 1 alpha C1D15: number analyzed (Participants) | 76 | 51
  MIP 1 alpha C1D15 | -1.842 (11.9129) | -0.320 (38.5273)
  MIP 1 alpha C2D1: number analyzed (Participants) | 76 | 46
  MIP 1 alpha C2D1 | -2.098 (12.0121) | -0.473 (35.4447)
  MIP 1 alpha C3D1: number analyzed (Participants) | 49 | 0
  MIP 1 alpha C3D1 | -1.167 (15.9038) |
  MIP 1 alpha V98: number analyzed (Participants) | 6 | 0
  MIP 1 alpha V98 | 7.563 (7.8802) |
  MIP 1 beta C1D15: number analyzed (Participants) | 78 | 70
  MIP 1 beta C1D15 | 0.032 (20.1490) | 5.746 (64.1386)
  MIP 1 beta C2D1: number analyzed (Participants) | 79 | 67
  MIP 1 beta C2D1 | -1.198 (31.4522) | 31.277 (261.3460)
  MIP 1 beta C3D1: number analyzed (Participants) | 50 | 0
  MIP 1 beta C3D1 | 1.850 (15.208) |
  MIP 1 beta V98: number analyzed (Participants) | 6 | 0
  MIP 1 beta V98 | 7.518 (11.9566) |
  PDGF AA 31 P1 C1D15: number analyzed (Participants) | 0 | 69
  PDGF AA 31 P1 C1D15 |  | -183.36 (2260.110)
  PDGF AA 31 P1 C2D1: number analyzed (Participants) | 0 | 66
  PDGF AA 31 P1 C2D1 |  | -268.83 (2054.666)
  PDGF AA 31 C3D1: number analyzed (Participants) | 0 | 0
  PDGF AA 31 V98: number analyzed (Participants) | 0 | 0
  PDGF AB C1D15: number analyzed (Participants) | 76 | 69
  PDGF AB C1D15 | -36.637 (353.6898) | -121.278 (325.1308)
  PDGF AB C2D1: number analyzed (Participants) | 77 | 66
  PDGF AB C2D1 | -99.852 (338.5816) | -80.778 (363.1249)
  PDGF AB C3D1: number analyzed (Participants) | 50 | 0
  PDGF AB C3D1 | -7.702 (311.6834) |
  PDGF AB V98: number analyzed (Participants) | 5 | 0
  PDGF AB V98 | 130.800 (382.6282) |
  PDGF BB C1D15: number analyzed (Participants) | 78 | 69
  PDGF BB C1D15 | -120.317 (1758.7655) | -567.664 (1385.6740)
  PDGF BB C2D1: number analyzed (Participants) | 79 | 66
  PDGF BB C2D1 | -435.311 (1961.7449) | -371.888 (1186.1)
  PDGF BB C3D1: number analyzed (Participants) | 51 | 0
  PDGF BB C3D1 | 333.637 (1516.1506) |
  PDGF BB V98: number analyzed (Participants) | 6 | 0
  PDGF BB V98 | 174.083 (3221.9009) |
  Placental Derived Growth Factor C1D15: number analyzed (Participants) | 78 | 56
  Placental Derived Growth Factor C1D15 | 55.444 (55.0671) | 55.0671 (29.8457)
  Placental Derived Growth Factor C2D1: number analyzed (Participants) | 79 | 54
  Placental Derived Growth Factor C2D1 | 50.439 (58.2571) | 51.359 (76.6390)
  Placental Derived Growth Factor C3D1: number analyzed (Participants) | 51 | 0
  Placental Derived Growth Factor C3D1 | 61.080 (58.2969) |
  Placental Derived Growth Factor V98: number analyzed (Participants) | 6 | 0
  Placental Derived Growth Factor V98 | 112.683 (110.3416) |
  Chemokine Ligand 5 C1D15: number analyzed (Participants) | 0 | 70
  Chemokine Ligand 5 C1D15 |  | -2373.94 (46225.695)
  Chemokine Ligand 5 C2D1: number analyzed (Participants) | 0 | 67
  Chemokine Ligand 5 C2D1 |  | 551.64 (49492.450)
  Chemokine ligand 5 C3D1: number analyzed (Participants) | 0 | 0
  Chemokine ligand 5 V98: number analyzed (Participants) | 0 | 0
  SDF 1 alpha C1D15: number analyzed (Participants) | 77 | 69
  SDF 1 alpha C1D15 | 441.305 (385.8988) | 506.768 (487.7603)
  SDF 1 alpha C2D1: number analyzed (Participants) | 77 | 66
  SDF 1 alpha C2D1 | 520.051 (510.8558) | 647.435 (470.0962)
  SDF 1 alpha C3D1: number analyzed (Participants) | 51 | 0
  SDF 1 alpha C3D1 | 509.483 (550.4383) |
  SDF 1 alpha V98: number analyzed (Participants) | 5 | 0
  SDF 1 alpha V98 | 836.532 (686.4434) |
  Soluble IL2 Receptor alpha C1D15: number analyzed (Participants) | 65 | 67
  Soluble IL2 Receptor alpha C1D15 | -25.869 (86.0991) | -414.669 (765.1544)
  Soluble IL2 Receptor alpha C2D1: number analyzed (Participants) | 67 | 64
  Soluble IL2 Receptor alpha C2D1 | -13.695 (65.5643) | -290.918 (1023.3392)
  Soluble IL2 Receptor alpha C3D1: number analyzed (Participants) | 41 | 0
  Soluble IL2 Receptor alpha C3D1 | -12.233 (31.5415) |
  Soluble IL2 Receptor alpha V98: number analyzed (Participants) | 4 | 0
  Soluble IL2 Receptor alpha V98 | -19.238 (43.0942) |
  TGF alpha C1D15: number analyzed (Participants) | 52 | 48
  TGF alpha C1D15 | -0.874 (4.6605) | 21.148 (168.7766)
  TGF alpha C2D1: number analyzed (Participants) | 51 | 43
  TGF alpha C2D1 | -0.350 (6.5375) | -6.019 (24.3258)
  TGF alpha C3D1: number analyzed (Participants) | 31 | 0
  TGF alpha C3D1 | 1.165 (11.8825) |
  TGF alpha V98: number analyzed (Participants) | 3 | 0
  TGF alpha V98 | 2.590 (3.4672) |
  Tie-2 C1D15: number analyzed (Participants) | 77 | 69
  Tie-2 C1D15 | -2971.948 (2397.5234) | -3573.856 (2996.7139)
  Tie-2 C2D1: number analyzed (Participants) | 78 | 66
  Tie-2 C2D1 | -3447.692 (3577.1791) | -4088.214 (3191.9812)
  Tie-2 C3D1: number analyzed (Participants) | 51 | 0
  Tie-2 C3D1 | -2811.765 (3459.1934) |
  Tie-2 V98: number analyzed (Participants) | 5 | 0
  Tie-2 V98 | -1924.000 (3215.5684) |
  TNF alpha C1D15: number analyzed (Participants) | 77 | 67
  TNF alpha C1D15 | -0.233 (4.9747) | 1.451 (24.8216)
  TNF alpha C2D1: number analyzed (Participants) | 78 | 64
  TNF alpha C2D1 | 0.039 (3.9540) | 1.741 (15.0677)
  TNF alpha C3D1: number analyzed (Participants) | 49 | 0
  TNF alpha C3D1 | 0.614 (4.6336) |
  TNF alpha V98: number analyzed (Participants) | 6 | 0
  TNF alpha V98 | 3.027 (4.7343) |
  VEGF C1D15: number analyzed (Participants) | 78 | 66
  VEGF C1D15 | -13.294 (112.6871) | 10.709 (285.2533)
  VEGF C2D1: number analyzed (Participants) | 78 | 62
  VEGF C2D1 | -11.523 (122.6064) | -26.215 (239.4960)
  VEGF C3D1: number analyzed (Participants) | 50 | 0
  VEGF C3D1 | 16.732 (160.3096) |
  VEGF V98: number analyzed (Participants) | 6 | 0
  VEGF V98 | 155.638 (352.8309) |
  VEGF A C1D15: number analyzed (Participants) | 78 | 69
  VEGF A C1D15 | 78.868 (174.8011) | 92.748 (273.6190)
  VEGF A C2D1: number analyzed (Participants) | 79 | 66
  VEGF A C2D1 | 76.041 (194.1394) | 140.664 (336.9135)
  VEGF A C3D1: number analyzed (Participants) | 51 | 0
  VEGF A C3D1 | 116.800 (233.1657) |
  VEGF A V98: number analyzed (Participants) | 6 | 0
  VEGF A V98 | 465.833 (515.7676) |
  VEGF D C1D15: number analyzed (Participants) | 78 | 21
  VEGF D C1D15 | 0.953 (87.6513) | 3.404 (42.7585)
  VEGF D C2D1: number analyzed (Participants) | 78 | 19
  VEGF D C2D1 | -9.776 (98.0905) | 11.043 (116.5445)
  VEGF D C3D1: number analyzed (Participants) | 51 | 0
  VEGF D C3D1 | 9.894 (57.1140) |
  VEGF D V98: number analyzed (Participants) | 6 | 0
  VEGF D V98 | -21.317 (88.6689) |
  VEGF Rec 1 C1D15: number analyzed (Participants) | 78 | 55
  VEGF Rec 1 C1D15 | 593.613 (3109.3343) | -221.867 (799.9202)
  VEGF Rec 1 C2D1: number analyzed (Participants) | 79 | 53
  VEGF Rec 1 C2D1 | -3.971 (739.7875) | -243.661 (1031.2376)
  VEGF Rec 1 C3D1: number analyzed (Participants) | 51 | 0
  VEGF Rec 1 C3D1 | -209.863 (809.7744) |
  VEGF Rec 1 V98: number analyzed (Participants) | 6 | 0
  VEGF Rec 1 V98 | -15.567 (90.6274) |
  VEGF Rec 2 C1D15: number analyzed (Participants) | 78 | 67
  VEGF Rec 2 C1D15 | -10110.096 (5626.0125) | -8842.040 (6078.7151)
  VEGF Rec 2 C2D1: number analyzed (Participants) | 78 | 64
  VEGF Rec 2 C2D1 | -9369.165 (17982.0625) | -10676.563 (7064.0825)
  VEGF Rec 2 C3D1: number analyzed (Participants) | 51 | 0
  VEGF Rec 2 C3D1 | -11389.576 (10955.1596) |
  VEGF Rec 2 V98: number analyzed (Participants) | 6 | 0
  VEGF Rec 2 V98 | -9021.217 (5921.9619) |
  VEGF Rec 3 C1D15: number analyzed (Participants) | 70 | 61
  VEGF Rec 3 C1D15 | -1174.650 (2226.7893) | -2251.867 (3231.1485)
  VEGF Rec 3 C2D1: number analyzed (Participants) | 68 | 58
  VEGF Rec 3 C2D1 | -1320.738 (3138.3810) | -2523.257 (3550.7291)
  VEGF Rec 3 C3D1: number analyzed (Participants) | 47 | 0
  VEGF Rec 3 C3D1 | -1488.140 (3687.8774) |
  VEGF Rec 3 V98: number analyzed (Participants) | 5 | 0
  VEGF Rec 3 V98 | -1201.680 (2441.5741) |

8. Secondary Outcome: Summary of Plasma Concentration of Lenvatinib
Description: Blood samples for the quantification of lenvatinib in plasma were obtained and processed using a standardized protocol. The lower limit of quantification was 0.25 ng/mL. Pharmacokinetic (PK) analysis was conducted using nonlinear mixed effects modeling. Descriptive statistics were used to summarize lenvatinib plasma concentration data.
Time Frame: Predose and 2 to 12 hours postdose at Cycle 1 Day 1 (C1D1), Cycle 1 Day 15 (C1D15), and Cycle 2 Day 1 (C2D1)
Population: The PK analysis set was used for analysis and included all participants who received at least one dose of lenvatinib and had at least one quantifiable lenvatinib concentration. Number analyzed (n) signifies participants who were evaluable at specific time points for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 (V600E BRAF Negative) | Cohort 2 (V600E BRAF Positive)
Number analyzed (Participants) | 93 | 89
ng/mL
  C1D1 Pre-dose: number analyzed (Participants) | 92 | 85
  C1D1 Pre-dose | 0 (0) | 0 (0)
  C1D1 Post-dose: number analyzed (Participants) | 89 | 85
  C1D1 Post-dose | 229.6 (148.98) | 287.6 (168.97)
  C1D15 Pre-dose: number analyzed (Participants) | 79 | 77
  C1D15 Pre-dose | 56.8 (82) | 71.9 (104.09)
  C1D15 Post-dose: number analyzed (Participants) | 80 | 79
  C1D15 Post-dose | 284.0 (141.71) | 332.1 (221.98)
  C2D1 Pre-dose: number analyzed (Participants) | 78 | 73
  C2D1 Pre-dose | 38.7 (32.94) | 52.0 (48.73)
  C2D1 Post-dose: number analyzed (Participants) | 74 | 68
  C2D1 Post-dose | 244.5 (182.67) | 270.4 (143.64)

ADVERSE EVENTS:
Time Frame: From date of administration of first dose up to 30 days after the last dose, or up to data cutoff (15 Jan 2012 and 15 Apr 2013 for Cohort 1 and Cohort 2, respectively), up to approximately 33 months.
Arm/Group | Cohort 1 (V600E BRAF Negative) | Cohort 2 (V600E BRAF Positive)
Serious Adverse Events (participants affected / at risk) | 39/93 | 36/89
Other Adverse Events (participants affected / at risk) | 93/93 | 88/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (V600E BRAF Negative) (N=93) | Cohort 2 (V600E BRAF Positive) (N=89)
Hypertension (Vascular disorders) | 5 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 3
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Oesophageal spasm (Gastrointestinal disorders) | 1 | 0
Rectal perforation (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 2
Appendicitis (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 1 | 0
Incision site infection (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Pelvic abscess (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Cranial nerve palsies multiple (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Urethral obstruction (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Atrial thrombosis (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mental status changes (Psychiatric disorders) | 2 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Gallbladder perforation (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Ejection fraction decreased (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 2
General physical health deterioration (General disorders) | 0 | 2
Impaired healing (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Chemical peritonitis (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (V600E BRAF Negative) (N=93) | Cohort 2 (V600E BRAF Positive) (N=89)
Anaemia (Blood and lymphatic system disorders) | 5 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 9
Hypothyroidism (Endocrine disorders) | 17 | 24
Abdominal pain (Gastrointestinal disorders) | 21 | 19
Abdominal pain upper (Gastrointestinal disorders) | 11 | 6
Constipation (Gastrointestinal disorders) | 25 | 28
Diarrhoea (Gastrointestinal disorders) | 44 | 26
Dry mouth (Gastrointestinal disorders) | 14 | 10
Dyspepsia (Gastrointestinal disorders) | 5 | 9
Flatulence (Gastrointestinal disorders) | 12 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 | 6
Glossodynia (Gastrointestinal disorders) | 6 | 2
Nausea (Gastrointestinal disorders) | 48 | 36
Oral pain (Gastrointestinal disorders) | 10 | 5
Stomatitis (Gastrointestinal disorders) | 16 | 12
Vomiting (Gastrointestinal disorders) | 36 | 32
Asthenia (General disorders) | 6 | 5
Chills (General disorders) | 6 | 4
Fatigue (General disorders) | 62 | 41
Oedema peripheral (General disorders) | 14 | 10
Pain (General disorders) | 6 | 5
Pyrexia (General disorders) | 7 | 10
Oral herpes (Infections and infestations) | 5 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 4
Urinary tract infection (Infections and infestations) | 10 | 9
Aspartate aminotransferase increased (Investigations) | 3 | 5
Blood alkaline phosphatase increased (Investigations) | 7 | 3
Blood thyroid stimulating hormone increased (Investigations) | 14 | 7
Gamma-glutamyltransferase increased (Investigations) | 5 | 1
Lipase increased (Investigations) | 7 | 3
Weight decreased (Investigations) | 22 | 12
Decreased appetite (Metabolism and nutrition disorders) | 40 | 30
Dehydration (Metabolism and nutrition disorders) | 6 | 12
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 8 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 12
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 8 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 6
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 7 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 13 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 | 9
Dizziness (Nervous system disorders) | 10 | 16
Dysgeusia (Nervous system disorders) | 12 | 16
Headache (Nervous system disorders) | 29 | 21
Lethargy (Nervous system disorders) | 1 | 5
Peripheral sensory neuropathy (Nervous system disorders) | 10 | 2
Confusional state (Psychiatric disorders) | 2 | 5
Depression (Psychiatric disorders) | 4 | 5
Insomnia (Psychiatric disorders) | 7 | 8
Haematuria (Renal and urinary disorders) | 5 | 3
Proteinuria (Renal and urinary disorders) | 23 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 11
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 26 | 33
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 16 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 5
Rash (Skin and subcutaneous tissue disorders) | 16 | 5
Hot flush (Vascular disorders) | 5 | 1
Hypertension (Vascular disorders) | 53 | 48
Hypotension (Vascular disorders) | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other